CLINICAL TRIAL: NCT06463600
Title: Tumour Localisation With Magnetic Clip Before Neoadjuvant Chemotherapy. A Randomised Pilot Feasibility Study: MagLocal 1.0
Brief Title: Tumour Localisation With Magnetic Clip Before Neoadjuvant Chemotherapy.
Acronym: MagLocal
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sahlgrenska University Hospital (Other)
Responsible Party: Principal Investigator, Professor Fredrik Warnberg, professor, Sahlgrenska University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SUGBG-2023001
Record Dates: First submitted 2024-06-11; First posted 2024-06-18 (Actual); Last update posted 2024-06-18 (Actual); Status verified 2024-06

CONDITIONS: Breast Conserving Surgery
Keywords: Breast cancer; Tumour localisation; Magnetic clip; magnetic tracer; Preoperative chemotherapy
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: One part feasibility and one part randomised.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Tumour localisation with Magseed (Experimental): Before preoperative chemotherapy a Magseed is inserted in the breast tumour
  Interventions: Device: Magseed
- Metallic marker + guide wire (Active Comparator): Before preoperative chemotherapy an ordinary metallic clip is inserted in the breast tumour. Before surgery a guide wire is inserted to localise the clip.
  Interventions: Device: Metallic clip and guide wire

INTERVENTIONS:
Device: Magseed — Tumour localizer
  Arms: Tumour localisation with Magseed
Device: Metallic clip and guide wire — Tumour localizers
  Arms: Metallic marker + guide wire

SUMMARY:
The feasibility of the use of magnetic clips for tumour localisation before preoperative chemotherapy in combination with superparamagnetic iron oxide nanoparticles (SPIO) as tracer for sentinel lymph node (SLN) detection and in combination with a magnetic clip in the index lymph node metastasis is studied.

DETAILED DESCRIPTION:
The overall aim is to demonstrate that the use of magnetic clips for tumour localisation before preoperative chemotherapy is feasible at breast cancer surgery and histopathological evaluation in combination with superparamagnetic iron oxide nanoparticles (SPIO) as tracer for sentinel lymph node (SLN) detection, and in combination with a magnetic clip in the index lymph node metastasis if targeted axillary surgery is planned.

ELIGIBILITY:
Inclusion Criteria:

1. Age above 18 years
2. Planned for preoperative chemotherapy before breast cancer surgery
3. Planned breast conserving surgery with targeted axillary dissection or sentinel lymph node biopsy using magnetic technique
4. SLN-biopsy with magnetic tracer or targeted axillary dissection using magnetic tracer and Magseed
5. Signed and dated written informed consent before the start of specific protocol procedures

Exclusion Criteria:

1. Pregnant or breast-feeding
2. Iron overload disease
3. Known hypersensitivity to iron or dextran compounds
4. Inability to understand given information and give informed consent or undergo study procedures
5. Planned MRI control for tumour response during chemotherapy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Breast conserving surgery
Enrollment: 44 (Estimated)
Dates: Start 2024-02-01 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Specimen volume | Perioperatively
  The surgical specimen is weighed after removal.

CONTACTS AND LOCATIONS:
Overall Officials: Roger Olofsson Bagge, prof, Principal Investigator — Sahlgrenska Academy at Gothenburg University
Locations (1):
- Sahlgrenska Academy at Gothenburg University, Gothenburg, Göteborg, Sweden

IPD SHARING:
Plan to Share IPD: No